CLINICAL TRIAL: NCT01989962
Title: Phase 2: Evaluation of Education for Equity (E4E)--Exploring How Health Professional Education Can Reduce Disparities in Chronic Disease Care and Improve Outcomes for Indigenous Populations
Brief Title: E4E-Health Professional Education for Improving Care for Canadian Aboriginal Populations
Acronym: E4E
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen's University (Other)
Collaborators: University of Calgary (Other); Laurentian University (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Michael Green, Associate Professor, Director for Centre for Health Services and Policy Research, Associate Director for Centre for Studies in Primary Care, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPID-439-13-E4E
Record Dates: First submitted 2013-10-15; First posted 2013-11-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus Type 2; Cultural Competency
Keywords: Aboriginal Health; Diabetes Mellitus Type 2; Cultural Competency; Continuing Medical Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E4E Intervention Group (Experimental): E4E Intervention Group is a group of family physicians who will participate in the first wave of E4E intervention.
  Interventions: Other: E4E intervention
- E4E Late Intervention Control Group (Sham Comparator): E4E Late Intervention Control Group is a group of family physicians who will participate in the second wave of E4E intervention 12 month later after the completion of the first wave of E4E intervention.
  Interventions: Other: E4E intervention

INTERVENTIONS:
Other: E4E intervention — The E4E intervention consists of a one-day face-to-face workshop and a series of follow-up online learning modules. Workshop and online content will be tailored to meet individual participants' needs determined by a pre-program needs assessment. E4E intervention will emphasize clinically based case scenarios and are designed to reinforce the workshop concepts and stimulate reflection. Participating family physicians will attend the workshop and engage in reflections and small-group interactions.
  Other Names: E4E continuing medical educational intervention

SUMMARY:
Education for Equity (E4E)intervention intends to improve care delivery through a well designed educational program that address not only the issues of diabetes care delivery to Aboriginal patients with diabetes, but also the issues of effective cross-cultural and culturally safe communication between healthcare providers and Aboriginal patients, and the issues related to effective implementation of appropriate chronic disease management programs for Aboriginal patients in a range of practice settings. The purpose of this study is to evaluate the effectiveness of the E4E education program through measuring patient clinical outcomes, patient experience with their doctors, and the changes in physicians' approaches to care perceived by Aboriginal diabetic patients.

DETAILED DESCRIPTION:
Two waves of the E4E intervention will be delivered to family physicians who have Aboriginal patients with type 2 diabetes on and off reserves. A mix-method approach will be employed in this evaluation study. Evaluation instruments include: (1) chart reviews and (2) patient experience surveys.

1. Chart review: A randomized, controlled, pre- and post intervention study design will be used to evaluate the effect of the E4E intervention on type 2 diabetes clinical outcomes of the Aboriginal patients. A retrospective chart audit will be used to gather the clinical data from 12 months prior to and 12 month after the intervention, not including the time during intervention.

   Sample Size for chart review: The primary outcome measure of HbA1C value will be used to identify the impact of E4E intervention on the clinical outcome of Aboriginal patients with type 2 diabetes. It is hypothesized that the A1C value would be reduced in the E4E Intervention Group's patients whose A1C values are at or above 8.0% prior to the E4E intervention (baseline) compared to the patients in E4E Late Intervention Control Group. A 0.5% difference of patients' A1C values between these two groups will be a clinically significant difference. The sample size needed to detect such a difference is estimated to be 98 eligible patients charts with A1C at or above 8.0% from E4E Intervention Group and 98 eligible patient charts from E4E Late Intervention Control Group, with an a=0.05 and ß=0.15. Given the proportion of 61.1% of Aboriginal patients with type 2 diabetes having A1C at or above 8.0%, we need to review 163 patient charts to obtain 98 eligible charts from each group. When 10 charts extractions per physician are performed, we need 17 physicians from each group. Considering a possible 20% loss to follow up, we need to recruit 20 physicians from E4E Intervention Group and 20 physicians from E4E Late Intervention Control Group, a total of 40 physicians to be invited to participate in chart reviews.

   Recruitment of physicians: After obtaining ethics approval from Queen's University Research Office, we will recruit 8-10 physicians to participate in the project at each potential site. Once recruitment is completed on each site, physicians will be randomized into E4E Intervention Group and E4E Late Intervention Control Group (sham comparator) who will participate in the second wave of E4E intervention 12 month later. Letters of information and consent form will be sent to the physicians to obtain their signed consent to participating in E4E chart review, patient survey and patient interview.

   Data collection regarding chart reviews for diabetes: The evaluation team will require the consenting physicians to create a list of all of their Aboriginal patients with type 2 diabetes using billing code 250, removing non-Aboriginal patients. This process can either be managed by the practice (with staff being reimbursed for time required) or can be conducted by the research staff at time of the chart audit. Each physician will then be asked to review the list for accuracy. Random number generation will be used to select charts at random from the list until the required number of eligible patient charts has been identified. Chart reviewers will be trained staff from the evaluation team and travel to each selected location to conduct chart audits.
2. Patient experience survey: Two (2) patient experience surveys will be conducted to evaluate the experience of Aboriginal patient with type 2 diabetes with his/her physician, respectively at the point of 3-month after the E4E intervention and at the point of 12-month after the intervention.

Sample size for patient experience surveys: An effective sample size needed for patient experience survey, with an a=0.05 and power 85% (ß=0.15), is estimated to be 102 eligible Aboriginal type 2 diabetic patients from E4E Intervention Group and the same number of eligible Aboriginal patients from E4E Late Intervention Control Group. We will recruit 10 eligible Aboriginal patients from each of the physicians in E4E Group A and 10 eligible Aboriginal patients from each of the physicians in E4E Group B. A total of 400 patients will be recruited to participate in Patient Experience surveys. This sample size (200 from each group) is more than sufficient to achieve 85% power even after allowing for drop out of physicians and any unanticipated difficulties in patient recruitment.

Data collection regarding patient experience surveys: The Patient Experience Surveys will take approximately 15-20 minutes to complete and will be completed on the day of patient visit. Patient Experience Survey is designed in two sections: pre-visit section and post visit section. Consent needs to be obtained from patients in pre-visit section.

* The receptionist of the selected practice will notify eligible patients about the study, and ask if they are willing to discuss with support/research staff about participating in a Patient Experience Survey. If the patient is interested, the receptionist will refer her/him to the onsite support/research staff, or provide access to a private phone with toll free number to contact support/research staff.
* Support/Research staff will review the information letter with the patient and obtain informed consent.
* The patient completes the pre-visit section and sign on the consent before seeing the doctor.
* After seeing the doctor, the patient will be asked to complete the post-visit survey and return it to the support/research staff before leaving the clinic. For patients who are not able to do so, they will be offered a choice to complete the survey by toll free telephone or fill in a hard copy of questionnaire and mail it out by pre-paid mail.
* Regular updates will be performed during data collection process to keep tack of patients participation in the survey.

ELIGIBILITY:
1. Family physicians Inclusion criteria

   * Fluent in English
   * Participate in the early or late E4E MAINPRO-C workshop
   * minimum 6 months in practice working with Aboriginal population
   * Minimum of 20 Aboriginal type 2 diabetic patients in patient roster
   * Intend to remain in practice location for 12 months post early intervention.

   Exclusion criteria:

   • Locum physician or plan to relocate before the study is completed
2. Patient chart inclusion criteria:

   Inclusion criteria
   * minimum 18 years of age
   * See the same physician for care over the course of study
   * minimum 5 years diagnosed with type 2 diabetes
   * Self identified as Aboriginal
   * A1C ≥ 8.0% at baseline (one year prior to the start of early E4E intervention)

   Exclusion criteria:
   * <18 years of age
   * Living in a nursing home
   * Physicians did not consent to audit
   * Type 1 diabetes or gestational diabetes diagnosis or impaired glucose
   * Not self-identified as Aboriginal population
   * A1C < 8.0% at baseline one year prior to intervention
3. Patients participating in Patient Experience Survey

Inclusion criteria:

* minimum 18 years of age
* See the same physician for care over the course of study
* minimum 5 years diagnosed with type 2 diabetes
* Self identified as Aboriginal
* Patients participating in interviews.

Exclusion criteria:

* <18 years of age
* Living in a nursing home
* Type 1 diabetes or gestational diabetes diagnosis or impaired glucose
* Not self-identified as Aboriginal population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C values--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  The primary outcome measure of A1C value will be used to identify the impact of the E4E program on clinical outcomes of Aboriginal patients with type 2 diabetes. It is hypothesized that the A1C value of the patients at or above 8.0% prior to their physicians' participation in the E4E intervention will be reduced since their physicians participate in the E4E intervention.
Cultural safety, bias and discrimination--change is being assessed | within 2 weeks after the E4E workshop; 1 year later after completetion of E4E intervention
  Physicians' cultural safety, bias and discrimination will be measured with a Cultural Competence, Sensitivity and Discrimination scale* from patients' perspectives. It is hypothesized that Aboriginal patients with type 2 diabetes will perceive increased cultural safety and decreased cultural bias/discrimination in their interactions with physicians since physicians participate in the E4E intervention.
  *Haggerty J, Burge F, Gass D, Santor D, Levesque JF, Beaulieu MD, Pineault R, Beninguisse G, Beauliur C. Evaluating the Quality of Primary Health Care from the Consumer Perspective: Validation of Instruments Adapted to the Canadian Context.(February 2006). Retrieved May 18th, 2013. Available at http://www.smhc.qc.ca/ignitionweb/data/media_centre_files/624/Mapping%20of%20PHC%20Attributes%20to%20Questionaries%20_%20final%20report%202006.pdf

SECONDARY OUTCOMES:
Diabetes process of care measures (date only)--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  Frequency of exams for complications of diabetes(eye, foot, ECG, waist circumference, neuropathy) is an indicator of quality of care related to physicians' adherence to diabetes care guidelines. It is hypothesized that the adherence to recommended screening for complications will be increased since physicians participate in the E4E intervention.
Other laboratory tests (values and date)--change is being assessed | a 12-month period prior to the start of the E4E intervention; a 12-month period after completion of the E4E intervention
  Frequency of other laboratory tests is an indicator of physicians' adherence to recommended control and prevention of complications. Test results are indicators of clinical outcomes of diabetes control in Aboriginal patients. The tests that will be examined are:
  1. Triglycerides
  2. HDL
  3. LDL
  4. Total cholesterol: HDL
  5. Total cholesterol
  6. eGFR/Creatinine Clearance
  7. Serum Creatinine
  8. A:C ratio
  9. 24 hour urine
  It is hypothesized that adherence to recommended tests and test results will be improved since physicians participate in the E4E intervention.
Blood pressure (systolic, diastolic, date)--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post completion of E4E intervention
  Frequency of blood pressure (BP) check is an indicator of physicians' adherence to recommended diabetes control and prevention of complications. BP values are an indicator of clinical outcome of diabetes control in Aboriginal patients with type 2 diabetes. It is hypothesized that physicians' adherence to recommended BP check and the BP results of Aboriginal patients with type 2 diabetes will be improved since physicians participate in the E4E intervention.
BMI (value, date)--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  Frequency of BMI check is an indicator of physicians' adherence to recommended diabetes control and prevention of complications. BMI values are an indicator of clinical outcomes of diabetes control in Aboriginal patients with type 2 diabetes. It is hypothesized that the adherence to BMI check will increased and BMI values will decrease since physicians participate in E4E intervention.
Medications--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post completion of E4E intervention
  Medications that physicians prescribe for their Aboriginal patients with type 2 diabetes will be examined, including:
  1. Anti-hyperglycemic medications
  2. Anti-hypertensive medications
  3. Lipid lowering medications
  4. Anti-coagulants (ASA, warfarin, etc.)
  It is hypothesized that the adherence to recommended control and prevention of complications will be increased since physicians participate in E4E intervention.
Diabetes counseling and education--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  Diabetes counseling and education that physicians provide to their Aboriginal patients with type 2 diabetes will be examined, including:
  1. exercises
  2. weight
  3. diet
  4. smoking cessation
  5. hypoglycemic event
  6. adjustment of treatment plan
  7. use of traditional medicine
  It is hypothesized that the adherence to recommended patient counseling and education will be increased since physicians participate in E4E intervention.
Documentation of self-management goals--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  Self-management goal is an indicator of efficacy of Aboriginal diabetic patients to self-management. It is hypothesized that Aboriginal patients with type 2 diabetes meet self-management goal better since their physicians participate in the E4E intervention.
Psychosocial self-efficacy scale of Aboriginal patients with type 2 diabetes (Diabetes Empowerment Scale Short Form)--change is being assessed | within 2 weeks after the E4E workshop; 1 year after the completion of E4E intervention
  Psychosocial self-efficacy scale of Aboriginal patients with type 2 diabetes will be examined through a Diabetes Empowerment Scale Short Form (DES SF)*. It is hypothesized that Aboriginal patients with type 2 diabetes will improve psychosocial self-efficacy since their physicians participate in the E4E intervention.
  * Anderson RM, Fitzgerald JT, Gruppen LD, Funnel MM, Oh MS. Diabetes Empowerment Scale Short Form (DSL SF). Diabetes Care 2003, 26(5):1641-2.
Patient experiences of healthcare service (Canadian Institute of Health Information (CIHI) Patient Experience Survey)--change is being assessed | within 2 weeks after the E4E workshop; 1 year later after the completion of E4E intervention
  Patients' healthcare experience will be assessed using the CIHI Patient Experience Survey* and the Diabetes Empowerment Scale Short Form immediately after the E4E workshops being delivered and one year after the workshops. A co-primary outcome is Summary Patient Experience Score. It is hypothesized that Aboriginal patients will have better healthcare experiences with their physicians who participated in the E4E intervention.
  * CIHI (2012). "Measuring Patient Experiences in Primary Health Care Survey". Retrieved September 10, 2013. Available at http://www.cihi.ca/CIHI-ext-portal/pdf/internet/INFO_PHC_PATIENT_EN

OTHER OUTCOMES:
Clinic visits--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  number of visits to healthcare providers is an indicator of adherence to control and prevention of complications. It is hypothesized that Aboriginal patients will increase visits to family physicians and allied healthcare providers (nurse, dietitian, social worker, pharmacist, diabetes nurse educator, traditional healer, etc.) since physicians participate in E4E intervention.
Referrals (to whom and date)--change is being assessed | a 12-month period prior to the start of E4E intervention; a 12-month period post the completion of E4E intervention
  Physician's referral of their Aboriginal patients with type 2 diabetes to other healthcare providers is an indicator of adherence to control and prevention of complications. It is hypothesized that since participating in E4E intervention, physicians will increase referral to a wider range of healthcare professionals such as diabetes specialist, diabetes education center (DEC), diabetes educator, pedorthist, chiropodist, optometrist, ophthalmologist, nephrologist, cardiology, EMG/Neurologist, dietician, urologist, internist, traditional healer, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Green, MD, Principal Investigator — Queen's University
Locations (1):
- Centre for Studies in Primary Care, Department of Family Medicine, Queen's University, Kingston, Ontario, Canada